CLINICAL TRIAL: NCT06023407
Title: Feasibility of Improving Glycemia With Heat Therapy to Prevent AD
Acronym: FIGHT-AD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00147285; R01AG081304 (NIH)
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy Aging; Alzheimer Disease; Metabolic Disease
MeSH Terms: conditions — Alzheimer Disease; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: 1:1 allocation to either heat therapy intervention or thermoneutral control group
Who Masked: Investigator
Masking Description: Primary Investigators will be blinded to participants group. Due to the type of intervention we are unable to blind participant or certain members of the study team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat therapy Group (Experimental): 40.5°C water
  Interventions: Other: Water Immersion Heat Therapy
- Thermoneutral Control Group (Sham Comparator): 36°C water
  Interventions: Other: Water Immersion Heat Therapy

INTERVENTIONS:
Other: Water Immersion Heat Therapy — 10-weeks of 3 days per week in 1 of the 2 arms

SUMMARY:
The investigators will determine if heat therapy can improve blood (Aim 1) and brain (Aim 2) glucose metabolism in cognitively healthy older adults (65+) who are at risk for AD. The investigators will also examine the degree to which changes in blood and brain glucose metabolism track together and explore several additional potential mechanisms that are critical to understanding the brain benefits of heat therapy (Aim 3). These aims will provide a comprehensive understanding of the impact of heat therapy on whole body metabolic function and brain health.

DETAILED DESCRIPTION:
Aim 1. Examine the effects of heat therapy on blood glucose regulation in older adults at risk for AD. The Investigators will determine the ability of 10 weeks of heat therapy (3 days/week) to improve blood glucose regulation in older adults at risk for AD. Our primary outcome measures will be change in glycated hemoglobin (HbA1c), and change in insulin sensitivity index (ISI) assessed pre- vs post-intervention. The Investigators will also perform continuous glucose monitoring for 7 days prior to and following the intervention, as well as monitor dietary patterns during the intervention. The Investigators hypothesize that 10 weeks of heat therapy will lower HbA1c values and improve ISI outcomes.

Aim 2. Test the effect of heat therapy on brain glucose metabolism. To date, no studies have examined the impact of heat therapy on brain glucose metabolism. Here The Investigators will determine the effect of 10 weeks of heat therapy on brain glucose metabolism in older adults at risk for AD. Our primary outcome measure will be change in [18F] fluorodeoxyglucose (FDG) global standardized uptake value ratio (SUVR) pre- vs post- heat therapy. The Investigators hypothesize that individuals will improve (increase) global cerebral glucose metabolism following 10 weeks of heat therapy. The Investigators further hypothesize that the degree of change in blood glucose metabolism will track with change in brain glucose metabolism.

Aim 3. Explore the effect of heat therapy on fluid biomarkers (proteostasis, inflammation, neuropathology) and neuroimaging markers of brain health. The Investigators will explore the effect of heat therapy on plasma markers of proteostasis (HSP's), inflammation (CRP, TNF, IL-6, JNK and IKK) and AD-related neuropathology (Amyloid/Tau/Neurodegeneration; A/T/N measures) markers in plasma at baseline and following 10 weeks of heat treatment. The Investigators will also obtain MRI measures of resting state metabolism, brain blood flow, and oxygen uptake for preliminary characterization of intervention-related changes. The Investigators hypothesize that proteostasis, inflammation, and AD neuropathology will be beneficially affected by heat treatment. The Investigators further hypothesize that the team will observe benefits in MRI-related brain outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Stable medication doses (>1 month)
* Post-menopausal
* Clinical Dementia Rating (CDR) of 0
* History of or current metabolic impairment (i.e. metabolic syndrome, pre-diabetes, Type 2 Diabetes, etc)

Exclusion Criteria:

* Excluded from or unable to complete an MRI scan. MRI compatible pacemakers will require cardiologist clearance prior to enrolling.
* ACSM Risk score stratification of "High" unless cleared by a physician prior to participation.
* Myocardial infarction or symptoms of coronary artery disease in the last 2 years.
* History of or current diagnosis of disorders with the potential to impair cognition (i.e. AD, Parkinson's disease, stroke (defined as clinical episode w/ neuroimaging evidence in appropriate area to explain symptoms)).
* Insulin-dependent (Type 1) Diabetes Mellitus.
* Clinically significant chronic disease such as cancer, HIV, or acquired immunodeficiency syndrome.
* Clinically significant depressive symptoms that may impair cognition, use of psychoactive and investigational medications, and significant visual or auditory impairment.
* Orthopedic complications that would preclude individuals from safely entering a hot tub.
* Untreated hypothyroidism or diseases associated with heat intolerance (i.e. Graves disease, etc).
* Contraindication for temperature pill ingestion (i.e. inflammatory bowel disease, diverticulitis or related).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
HbA1C | 10 weeks
  hemoglobin A1C (HbA1C) test is a blood test that shows what your average blood sugar (glucose) level was over the past two to three months. below 5.7 %. Anyone with an HbA1c. A value of 5.7 % to 6.4 % is considered to be prediabetic, while diabetes can be diagnosed with a HbA1c of 6.5% or higher.
Insulin sensitivity index | 10 weeks
  Using glucose and insulin from a the OGTT, an indices will be calculated for insulin sensitivity. The goal is to increase the insulin sensitivity. Minimum=0; No upper limit. Increasing value indicates improved outcomes.

SECONDARY OUTCOMES:
Fluorodeoxyglucose (FDG) positron emission tomography (PET) Metabolism (Standard Uptake Value Ratio) | 10 weeks
  FDG PET measures reflecting cerebral metabolism standardized to the uptake value of the cerebellum and standardized uptake value ratios (SUVR) will be calculated from native-space region of interest (ROI).

CONTACTS AND LOCATIONS:
Overall Officials: Jill Morris, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Univeristy of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geiger PC, Pennington JS, Kueck PJ, John CS, Mayfield HD, Kemna RE, Burns J, Vidoni E, Honea R, Li Y, Mahnken J, Morris JK. Heat therapy in individuals at risk for Alzheimer's disease-methods for a randomized controlled trial. Front Neurol. 2026 Jan 23;17:1736108. doi: 10.3389/fneur.2026.1736108. eCollection 2026. PMID 41657418